CLINICAL TRIAL: NCT00916773
Title: Exercised-Induced Bronchoconstriction in Patients With Severe Obstructive Sleep Apnea
Brief Title: Pulmonary Disorders During Exercise in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Liying Wang, School and Graduate Institute of Physical Therapy, National Taiwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200712118R
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Sleep Apnea, Obstructive; Asthma, Exercise-Induced
Keywords: Obstructive sleep apnea; Airway inflammation; Exercise-induced bronchoconstriction; Continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Asthma, Exercise-Induced | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — CPAP of optimal pressure used during sleep for 3 months

SUMMARY:
Purposes:

1. To investigate whether patients with severe obstructive sleep apnea syndrome (OSAS) are at higher risk for exercised-induced bronchoconstriction (EIB) due to baseline airway inflammation compared with age, gender, and body mass index (BMI)-matched controls.
2. To investigate the effect of 3-month continuous positive airway pressure (CPAP) therapy on EIB for patients with severe OSAS.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized by repeated episodes of upper airway obstruction during sleep. Recent studies have found evidence of airway inflammation in patients with OSAS. Individuals with chronic airway inflammation are at higher risk for exercise-induced bronchoconstriction (EIB). We hypothesized patients with OSAS are at higher risk for EIB due to baseline airway inflammation. Continuous positive airway pressure (CPAP) is a known standard treatment for OSAS, thus the second aim of the study will be investigating the effect of 3-month CPAP therapy on EIB for patients with OSAS. Twenty severe OSAS patients and 20 control individuals matched for age, gender, and body mass index (BMI) will be recruited. All participants will come to the laboratory on 2 separate days (5~14 days interval). On the 1st visit, baseline pulmonary function test (PFT) and airway inflammation assess by induced sputum will be performed. On the 2nd visit, an exercise challenge test will be performed using standard testing protocol and post-exercise forced expiratory volume in one second (FEV1) will be measured at 2.5, 5, 10, 15,20, and 30 minutes. For patients with severe OSAS, all measurements will be repeated after 3-month CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged 18-65 y/o
2. Severe OSA (AHI≧30/hr)
3. BMI<35 kg/m2

Exclusion Criteria:

1. Clinical asthma
2. Chronic lung disease (FEV1<70% predicted or FEV1/FVC<70%)
3. Exercise contraindication:

   * Stroke or heart attack in last 3 months
   * Major cardiovascular disease
   * Unstable angina
   * Unable to perform cycle ergometry due to musculoskeletal problems
4. Respiratory tract infection in the past 2 weeks
5. Inability to perform acceptable-quality spirometry
6. Refuse to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of changed forced expiratory volume in 1 second. (to determine if an exercise-induced bronchoconstriction attacked) | 3 month

SECONDARY OUTCOMES:
Percentage of different inflammatory cells in induced sputum. (to determine to severity of baseline airway inflammation) | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Liying Wang, Ph.D., Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan